CLINICAL TRIAL: NCT00246675
Title: Frusemide Infusion for the Prevention of Deterioration of Renal Function in Post Cardiac Surgery
Brief Title: Frusemide Infusion for the Prevention of Deterioration in Renal Function Post Cardiac Surgery.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has ceased recruiting as Ethics approval has lapsed and the investigator availability reduced.
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2002.167
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Renal Impairment After Cardiac Surgery
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): Patients will only receive frusemide as per the treating physicians treatment
  Interventions: Drug: Frusemide
- Intervention (Other): Patients will be given frusemide to achieve a study specified urine output target of 1-2mls/kg/hour
  Interventions: Drug: Frusemide

INTERVENTIONS:
Drug: Frusemide

SUMMARY:
The purpose of the project is to test whether or not the commonly used medication frusemide, given after heart surgery, and aiming to increase urinary output can have an effect on kidney function.

DETAILED DESCRIPTION:
All patients will receive standard supportive care based on current established management practice of cardio-thoracic patients. The only difference in treatment will be the randomisation of patients to receive/not receive protocolised administration of frusemide targeting a urine output.

There will be 2 groups of patients. The control group-which will receive frusemide bolus doses if required as determined by the surgeon/consultant physician. The frusemide infusion group-which will be monitored to achieve a trial specified hourly urine output target range of 1-2mls/kg/hour. In order to achieve this target the patient may need to receive a loading dose of frusemide and may also then require a frusemide infusion. The aim will be to maintain the urine output within the target range for the first 48 hours after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted for cardiac surgery will be assessed for eligibility. Participants will be approached for inclusion, from the pre-admission clinics and wards of the Cardiothoracic surgery unit. Potential participants will be identified by the daily review of planned cardiothoracic surgery schedule.

Exclusion Criteria:

1. Already in established dialysis dependent chronic renal failure.
2. Known allergy to frusemide
3. Age < 18 years
4. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The incidence of increase in creatinine of 0.05 mmol/L or greater in the first 72 hours after cardiac surgery.

SECONDARY OUTCOMES:
1. The maximum change in serum creatinine from baseline value during the first 7 days of hospital stay.
2. Incidence of renal failure requiring any form of renal replacement therapy.
3. Duration of post-operative hospital and ICU stay.
4. The maximum Sequential Organ Failure Assessment (SOFA) score in the first 7 days of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: John F Cade, Principal Investigator — Royal Melbourne Hospital, Intensive Care Unit
Locations (1):
- Intensive Care Unit, Royal Melbourne Hospital, Parkville, Victoria, Australia